CLINICAL TRIAL: NCT00687284
Title: Observational Study on Evaluation of Glycaemic Control in Patients Using Levemir® (Insulin Detemir) as Initiation Insulin Therapy by Levemir® (Insulin Detemir) Administered Once Daily as the Treatment for Type 2 Diabetes Mellitus.
Brief Title: Observational Study of Glycaemic Control in Patients Uncontrolled on Oral Antidiabetic Agents and Starting With 1 (Once) Daily Levemir® (Insulin Detemir) as the Treatment of Type 2 Diabetes Mellitus
Acronym: START
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3515
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: Levemir®

SUMMARY:
This study is conducted in Europe. An observational study evaluating glycaemic control in patients using Levemir® as initiation insulin therapy as the treatment of type 2 diabetes in Slovakia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Patients inadequately controlled by OAD
* Patients willing to sign informed consent
* Selection of study participants at the discretion of the physician
* Particular attention should be paid to the drug interactions that are listed within the product label

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for the final visit;
* Subjects who were previously enrolled in this study
* Subjects with a hypersensitivity to insulin detemir or to any of the excipients.
* Women who are pregnant, breastfeeding or have the intention of becoming pregnant within next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetes mellitus type 2
Sampling Method: Non-Probability Sample
Enrollment: 2188 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in glycaemic control as measured by HbA1c. | For the duration of the study

SECONDARY OUTCOMES:
Percentage of subjects to reach HbA1c below 7.0% and below or equal 6.5% | After 12 weeks and 24 weeks
The effect on glycaemic control as measured by FPG | After 12 weeks and 24 weeks
Change in body weight | After 12 weeks and 24 weeks
Change in waist and hip perimeter | After 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Košice, Slovakia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com